CLINICAL TRIAL: NCT02062502
Title: A Phase III Double Blind, Randomized, Multicenter, Controlled Study to Evaluate the Immunogenicity, Safety, and Tolerability of VARIVAX™ New Seed Process (NSP) Administered Concomitantly With M-M-R™ II
Brief Title: Evaluation of Immunogenicity and Safety of VARIVAX™ New Seed Process (NSP) in Children (V210-063)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: V210-063
Record Dates: First submitted 2014-02-12; First posted 2014-02-13 (Estimated); Results first posted 2016-03-01 (Estimated); Last update posted 2018-10-30 (Actual); Status verified 2018-10

CONDITIONS: Varicella
MeSH Terms: conditions — Chickenpox | interventions — Measles-Mumps-Rubella Vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- VARIVAX™ NSP + M-M-R II™ (Experimental): VARIVAX™ New Seed Process 0.5 mL administered in the left arm and M-M-R II™ vaccine 0.5 mL administered in the right arm by subcutaneous injection on Day 1 and Day 91
  Interventions: Biological: VARIVAX™ New Seed Process; Biological: M-M-R II™
- VARIVAX™ 2007 Process + M-M-R II™ (Active Comparator): VARIVAX™ 2007 Process 0.5 mL administered in the left arm and M-M-R II™ vaccine 0.5 mL administered in the right arm by subcutaneous injection on Day 1 and Day 91
  Interventions: Biological: VARIVAX™ 2007 process; Biological: M-M-R II™

INTERVENTIONS:
Biological: VARIVAX™ New Seed Process — Varicella virus vaccine live manufactured with a new seed process
  Arms: VARIVAX™ NSP + M-M-R II™
Biological: VARIVAX™ 2007 process — Varicella virus vaccine live manufactured with the 2007 process
  Arms: VARIVAX™ 2007 Process + M-M-R II™
Biological: M-M-R II™ — Measles, Mumps, and Rubella virus vaccine live

SUMMARY:
This study will evaluate the immunogenicity, safety, and tolerability of VARIVAX™ (Varicella Virus Vaccine Live) manufactured with a New Seed Process (NSP) compared with the VARIVAX™ 2007 process. The primary hypotheses being tested are that antibody response rate and mean antibody titer induced at 6 weeks after a single vaccination by VARIVAX™ NSP are non-inferior to those induced by VARIVAX™ 2007 process, and that antibody response rate induced by VARIVAX™ NSP is acceptable.

ELIGIBILITY:
Inclusion Criteria:

* Negative clinical history for varicella, herpes zoster, measles, mumps, and rubella

Exclusion Criteria:

* Received any measles, mumps, rubella, or varicella vaccine at any time prior to the study, or is anticipated to receive any of these vaccines outside the study
* Any congenital or acquired immune deficiency, neoplastic disease, or depressed immunity
* Received systemic immunomodulatory steroids within 3 months prior to entering the study or is expected to receive them during the course of the study
* History of allergy or anaphylactic reaction to neomycin, gelatin, sorbitol, egg proteins, chicken proteins, or any component of VARIVAX™ or M-M-R II™
* Received salicylates within 14 days prior to study vaccination
* Exposed to varicella, herpes zoster, measles, mumps, or rubella in the 4 weeks prior to study vaccination
* Received immune globulin, a blood transfusion, or blood-derived products within 5 months prior to study vaccination
* History of seizure disorder, including febrile seizure
* Fever illness (>=102.2 °F [39.0 °C] within 72 hours prior to study vaccination
* History of thrombocytopenia
* Born to a human immunodeficiency virus (HIV)-infected mother
* Participated in any other clinical trial (other than a surveillance study) within 30 days prior to study enrollment.

Ages: 12 Months to 23 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 611 (Actual)
Dates: Start 2014-03-07 (Actual); Primary Completion 2015-02-24 (Actual); Study Completion 2015-10-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Senders SD, Bundick ND, Li J, Zecca C, Helmond FA. Evaluation of immunogenicity and safety of VARIVAX New Seed Process (NSP) in children. Hum Vaccin Immunother. 2018 Feb 1;14(2):442-449. doi: 10.1080/21645515.2017.1388479. Epub 2017 Dec 11. PMID 29087781

RESULTS

PARTICIPANT FLOW:
Groups:
- VARIVAX™ New Seed Process + M-M-R II™: VARIVAX™ New Seed Process 0.5 mL administered in the left arm and M-M-R II™ vaccine 0.5 mL administered in the right arm by subcutaneous injection on Day 1 and Day 91.
Period: Overall Study
Arm/Group | VARIVAX™ New Seed Process + M-M-R II™ | VARIVAX™ 2007 Process + M-M-R II™
Started | 306 | 305
Vaccinated Dose 1 | 306 | 305
Completed | 263 | 270
Not Completed | 43 | 35

BASELINE CHARACTERISTICS:
Population: All randomized participants
Groups:
- Total: Total of all reporting groups
Arm/Group | VARIVAX™ New Seed Process + M-M-R II™ | VARIVAX™ 2007 Process + M-M-R II™ | Total
Number analyzed (Participants) | 306 | 305 | 611
Age, Continuous [Mean (Standard Deviation); unit: Months] | 12.9 (1.9) | 12.8 (1.7) | 12.9 (1.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 140 | 139 | 279
  Male | 166 | 166 | 332

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Varicella Zoster Virus (VZV) Antibody Levels >=5 Glycoprotein Enzyme-linked Immunosorbent Assay (gpELISA) Units/mL
Time Frame: 6 weeks (43 days) after vaccination 1
Population: The analysis population is participants with a seronegative antibody titer at baseline and postvaccination serology contributing to the per-protocol analysis.
Measure: Number; unit: Percentage of participants
Arm/Group | VARIVAX™ New Seed Process + M-M-R II™ | VARIVAX™ 2007 Process + M-M-R II™
Number analyzed (Participants) | 254 | 254
Percentage of participants | 97.2 | 97.2
Statistical Analysis 1: Comparison: VARIVAX™ New Seed Process + M-M-R II™ vs VARIVAX™ 2007 Process + M-M-R II™; Test type: Non-Inferiority or Equivalence — The conclusion of non-inferiority (similarity) is based on the lower bound of the 2-sided 95% CI on the risk difference excluding a decrease equal to or more than the prespecified criterion of 10.0 percentage points for Varicella zoster virus; p < 0.001, Miettinen and Nurminen; Risk Difference (RD) = 0.0, 95% CI 2-sided [-3.2 to 3.2]

2. Primary Outcome: Geometric Mean Titer of VZV Antibodies
Description: Antibody titers were measured with gpELISA.
Time Frame: 6 weeks (43 days) after vaccination 1
Population: The analysis population is participants with seronegative antibody titer at baseline and postvaccination serology contributing to the per-protocol analysis.
Measure: Geometric Mean (95% Confidence Interval); unit: gpELISA units/mL
Arm/Group | VARIVAX™ New Seed Process + M-M-R II™ | VARIVAX™ 2007 Process + M-M-R II™
Number analyzed (Participants) | 254 | 254
gpELISA units/mL | 16.28 [15.11 to 17.55] | 17.2 [15.86 to 18.65]
Statistical Analysis 1: Comparison: VARIVAX™ New Seed Process + M-M-R II™ vs VARIVAX™ 2007 Process + M-M-R II™; Test type: Non-Inferiority or Equivalence — The conclusion of non-inferiority (similarity) is based on the lower bound of the 2-sided 95% CI on fold-difference, excluding a decrease of 1.5 fold or more; p < 0.001, t-test, 2 sided; Risk Difference (RD) = 0.95, 95% CI 2-sided [0.85 to 1.06]
Statistical Analysis 2: Comparison: VARIVAX™ New Seed Process + M-M-R II™; The conclusion of acceptability is based on the lower bound of the 95% Confidence Interval (CI) being >76%, and implies that the value of the parameter is statistically significantly greater than the prespecified acceptability criterion (76%); Test type: Superiority or Other; p < 0.001, Exact CI method/binomial proportion; Antibody Response Rate = 97.2, 95% CI 2-sided [94.4 to 98.9]

3. Secondary Outcome: Percentage of Participants With Fever (>=102.2 °F Oral Equivalent)
Time Frame: Up to 42 days after Vaccination 1 and Vaccination 2 (up to 133 days)
Population: The analysis population is All Subjects as Treated with temperature data at the time of assessment.
Measure: Number; unit: Percentage of participants
Arm/Group | VARIVAX™ New Seed Process + M-M-R II™ | VARIVAX™ 2007 Process + M-M-R II™
Number analyzed (Participants) | 291 | 293
Percentage of participants
  Up to 42 days after Vaccination 1: n=285, 287 | 9.5 | 10.5
  Up to 42 days after Vaccination 2: n=258, 267 | 8.1 | 8.6

4. Secondary Outcome: Percentage of Participants With Systemic Measles-like, Rubella-like, Varicella-like Rash, Mumps-like Symptoms, and Injection-site Rash After Vaccination 1
Time Frame: Up to 42 days after Vaccination 1
Population: The analysis population is All Subjects as Treated with results after Vaccination 1.
Measure: Number; unit: Percentage of participants
Arm/Group | VARIVAX™ New Seed Process + M-M-R II™ | VARIVAX™ 2007 Process + M-M-R II™
Number analyzed (Participants) | 291 | 293
Percentage of participants
  Measles-like Rash | 0.3 | 2.4
  Rubella-like Rash | 0.0 | 0.0
  Varicella-like Rash | 0.0 | 0.3
  Mumps-like Symptoms | 0.0 | 0.0
  Injection-site Rash | 0.3 | 1.4

5. Secondary Outcome: Percentage of Participants With Systemic Measles-like, Rubella-like, Varicella-like Rash, Mumps-like Symptoms, and Injection-site Rash After Vaccination 2
Time Frame: Up to 42 days after Vaccination 2
Population: The analysis population is All Subjects as Treated with results after vaccination 2
Measure: Number; unit: Percentage of participants
Arm/Group | VARIVAX™ New Seed Process + M-M-R II™ | VARIVAX™ 2007 Process + M-M-R II™
Number analyzed (Participants) | 277 | 276
Percentage of participants
  Measles-like Rash | 0.0 | 0.0
  Rubella-like Rash | 0.0 | 0.0
  Varicella-like Rash | 0.4 | 0.0
  Mumps-like Symptoms | 0.0 | 0.0
  Injection-site Rash | 0.7 | 0.0

6. Secondary Outcome: Percentage of Participants With Solicited Injection-site Erythema, Injection-site Swelling, and Injection-site Pain/Tenderness After Vaccination 1
Time Frame: Up to 5 days after Vaccination 1
Population: The analysis population is All Subjects as Treated with results after Vaccination 1.
Measure: Number; unit: Percentage of participants
Arm/Group | VARIVAX™ New Seed Process + M-M-R II™ | VARIVAX™ 2007 Process + M-M-R II™
Number analyzed (Participants) | 291 | 293
Percentage of participants
  Injection-site Erythema | 20.3 | 19.8
  Injection-site Swelling | 10.0 | 10.6
  Injection-site Pain/Tenderness | 29.9 | 28.0

7. Secondary Outcome: Percentage of Participants With Solicited Injection-site Erythema, Injection-site Swelling, and Injection-site Pain/Tenderness After Vaccination 2
Time Frame: Up to 5 days after Vaccination 2
Population: The analysis population is All Subjects as Treated with results after vaccination 2.
Measure: Number; unit: Percentage of participants
Arm/Group | VARIVAX™ New Seed Process + M-M-R II™ | VARIVAX™ 2007 Process + M-M-R II™
Number analyzed (Participants) | 277 | 276
Percentage of participants
  Injection-site Erythema | 20.6 | 22.5
  Injection-site Swelling | 16.2 | 12.0
  Injection-site Pain/Tenderness | 22.4 | 24.3

ADVERSE EVENTS:
Time Frame: SAEs: up to Day 271; Other AEs: up to 42 days after vaccination 1 or 2, injection-site AEs up to 5 days after vaccination 1 or 2
Description: The at-risk safety population is All Subjects as Treated with safety results.
Arm/Group | VARIVAX™ New Seed Process + M-M-R II™ | VARIVAX™ 2007 Process + M-M-R II™
Serious Adverse Events (participants affected / at risk) | 6/291 | 9/293
Other Adverse Events (participants affected / at risk) | 225/291 | 224/293
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VARIVAX™ New Seed Process + M-M-R II™ (N=291) | VARIVAX™ 2007 Process + M-M-R II™ (N=293)
Drowning (General disorders) | 0 (0) | 1 (1)
Bronchiolitis (Infections and infestations) | 0 (0) | 3 (3)
Gastroenteritis (Infections and infestations) | 2 (2) | 0 (0)
Groin abscess (Infections and infestations) | 0 (0) | 1 (1)
Lobar pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Otitis media acute (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 2 (2) | 1 (1)
Staphylococcal infection (Infections and infestations) | 0 (0) | 1 (1)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Status asthmaticus (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VARIVAX™ New Seed Process + M-M-R II™ (N=291) | VARIVAX™ 2007 Process + M-M-R II™ (N=293)
Diarrhoea (Gastrointestinal disorders) | 37 (42) | 22 (25)
Vomiting (Gastrointestinal disorders) | 28 (34) | 18 (21)
Injection site erythema (General disorders) | 95 (181) | 94 (190)
Injection site pain (General disorders) | 106 (272) | 117 (270)
Injection site swelling (General disorders) | 61 (110) | 59 (96)
Pyrexia (General disorders) | 60 (86) | 60 (87)
Conjunctivitis (Infections and infestations) | 12 (12) | 15 (15)
Otitis media (Infections and infestations) | 35 (38) | 33 (36)
Otitis media acute (Infections and infestations) | 23 (24) | 14 (16)
Upper respiratory tract infection (Infections and infestations) | 46 (59) | 44 (51)
Viral rash (Infections and infestations) | 6 (6) | 17 (18)
Irritability (Psychiatric disorders) | 17 (18) | 13 (18)
Cough (Respiratory, thoracic and mediastinal disorders) | 18 (20) | 25 (29)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 17 (18)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 31 (37) | 26 (35)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 25 (28) | 27 (30)
Rash (Skin and subcutaneous tissue disorders) | 23 (27) | 14 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results.